CLINICAL TRIAL: NCT02433951
Title: Exercise Tolerance in Patients With Coronary Artery Bypass Surgery (CABG) and Sternotomy vs. Patients With Minimally Invasive Coronary Surgery
Brief Title: Exercise Tolerance in Patients With CABG and Sternotomy vs. Patients With Minimally Invasive Coronary Surgery
Acronym: ENDO-ACAB
Status: Completed | Type: Observational
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Dominique Hansen, Associate professor, Hasselt University
Other Study IDs: ENDO-ACAB study
Record Dates: First submitted 2015-04-24; First posted 2015-05-05 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Coronary Artery Bypass Surgery
Keywords: exercise tolerance
MeSH Terms: interventions — Exercise Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- healthy individuals: Age, gender and BMI matched healthy subjects without any chronic disease or physical disability, and being sedentary.
  Interventions: Other: Cardiopulmonary exercise test
- CABG patients: Age, gender and BMI matched CABG patients, without neurologic, nephrologic, respiratory disease.
  Interventions: Other: Cardiopulmonary exercise test
- endo-ACAB patients: Age, gender and BMI matched endo-ACAB patients without neurologic, nephrologic, respiratory disease.
  Interventions: Other: Cardiopulmonary exercise test

INTERVENTIONS:
Other: Cardiopulmonary exercise test — Maximal exercise test with ergospirometry.

SUMMARY:
In this study, up to 20 healthy individuals, 20 endo-ACAB patients, and 20 CABG patients undergo a maximal cardiopulmonary exercise test after hospital discharge (for patients only). Exercise tolerance is compared between groups.

DETAILED DESCRIPTION:
In this prospective observational study, up to 20 healthy individuals (no history or presence of any chronic disease, sedentary), 20 endo-ACAB patients, and 20 CABG patients (matched for age, gender and BMI) undergo a maximal cardiopulmonary exercise test after hospital discharge (for patients only).During this exercise test, following parameters are assessed at peak effort and at the second ventilatory threshold (determined by VE/VCO2 slope method): oxygen uptake (VO2), oxygen saturation (SaO2), carbon dioxide output (VCO2), resoiratory gas exchange ratio (RER), expiratory volume (VE), ventilatory equivalent for VCO2 (VE/VCO2), ventilatory equivalent for VO2 (VE/VO2), end-tidal O2 pressure (PETO2), end-tidal CO2 pressure (PETCO2), heart rate (HR), oxygen pulse (VO2/HR), cycling power output (W), tidal volume (Vt), respiratory rate (RR), systolic blood pressure (SBP), diastolic blood pressure (DBP), rate pressure product (RPP). Peak exercise effort is validated by RERpeak.

ELIGIBILITY:
Inclusion Criteria:

* undergoing this type of surgery. For healthy subjects: must be sedentary.

Exclusion Criteria:

* any neurologic, nephrologic, respiratory disease. For healthy subjects: any chronic disease or condition.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing CABG surgery or endo-ACAB surgery.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2015-02; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
VO2peak (peak oxygen uptake) | At peak exercise, single measurement which is executed between 2-4 weeks after surgery.
  Peak oxygen uptake capacity, expressed as ml/min.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Dendale, Study Director — Jessa Hospital, Stadsomvaart 11, 3500 Hasselt, Belgium
Locations (1):
- Jessa Hospital, Hasselt, Belgium